CLINICAL TRIAL: NCT06373198
Title: Implementation of a Re-engagement Program for Hepatitis C Patients Lost to Follow-up in Argentina.
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital El Cruce (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Fernando Mario Cairo, Principal Investigator, Hospital El Cruce
Other Study IDs: 0040/2023-versión 1.0
Record Dates: First submitted 2024-02-22; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Hepatitis C Chronic; Hepatitis C
Keywords: viral hepatitis; treatment; direct antivirals agents; relink; linkage to care
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- i. Strategy to re-engage HCV patients in a high complex hospital with a network: An evaluation of the positivity of the hepatitis C test will be carried out. Positive patients will be included in the follow-up and specific treatment will be requested to achieve a cure. Standard of care will be applied.
  Interventions: Other: standard of care

INTERVENTIONS:
Other: standard of care — An evaluation of the positivity of the hepatitis C test will be carried out. Positive patients will be included in the follow-up and specific treatment will be requested to achieve a cure. Standard of care will be applied.

SUMMARY:
Hepatitis C virus (HCV) is a leading cause of morbidity and mortality worldwide. This infection continues to represent a major global public health concern. This is why the introduction of potent antivirals for the treatment of HCV has been one of the major breakthroughs of the current medical era.

From a public health perspective, HCV prevalence will be eliminated if the available treatment also targets those most likely to transmit the virus. Despite this scientific advance, a systematic review from the U.S. described that of the 43% of patients aware of their HCV diagnosis, only 16% started treatment. Clearly, the long-known barriers to accessing this treatment must be broken down in order to administer these effective antivirals. The World Health Organization (WHO) has set the ambitious goal of eliminating viral hepatitis as a public health threat by 2030. This goal is really difficult to achieve, especially in low and middle-income countries. Particularly in Argentina, there is a need to improve diagnosis, access to care, and treatment of viral hepatitis. The prospect of viral hepatitis elimination in our country is daunting due to the complexity of the health system and the cost of implementing different strategies. The most pragmatic approach would be to break down national elimination targets into smaller targets for individual populations, for which treatment and prevention interventions can be delivered more quickly and efficiently. This concept is known as micro-elimination. Focusing on micro-elimination of viral hepatitis means working to achieve the WHO target in specific subpopulations. Subpopulations known to have a higher prevalence of HCV infection include prisoners, people who inject drugs, and patients requiring hemodialysis, among others.

Currently, patient unawareness of HCV infection represents one of the major barriers to treatment. In many cases, the diagnosis of HCV was established many years ago and patients do not seek treatment probably because they do not recognize the urgency of treating this asymptomatic infection. It is our goal, then, to identify the group of individuals who have been diagnosed with HCV infection but are not currently undergoing regular visits with health care professionals. This strategy is now called re-linking to the medical care of patients with chronic HCV.

DETAILED DESCRIPTION:
The protocol consists of implementing a strategy to contact patients with HCV who have been lost to follow-up. Establish a single model of confidential information management.

Population. From a cohort of patients, a non-probabilistic sampling of subjects meeting the eligibility criteria will be performed

Study Variables - Demographic data: age, gender

HCV-related data:

* Hepatic complications such as hepatocarcinoma, ascites, encephalopathy, variceal hemorrhage and liver transplantation.
* Extrahepatic manifestations such as non-Hodgkin's lymphoma, cryoglobulinemia, porphyria cutanea tarda, cardiovascular disease, diabetes mellitus.
* Previous antiviral treatment with interferon-based or direct antiviral drugs.

Sources of information

* Patient contact: phone call and/or e-mail.
* Review of electronic medical records.

Patient contact strategy:

- Patients identified as lost to follow-up will be contacted by telephone. Initially 3 calls will be made from Monday to Friday. If the patient is not located, he/she will be called on a Saturday and an e-mail will be sent (if available).

Possible outcomes after the intervention:

* Not contacted despite implemented strategy
* Death
* Treated at another center
* Contacted and candidate for follow-up

Measurement and data logging:

A specific form will be used to record the data, which will later be entered into a computerized database for subsequent analysis of the information. The research physicians who will be blinded will collect the exposure variables included in the survey to the results. Data for each patient will be obtained from the computerized medical record. Those patients with chronic HCV and whose disease course is unknown will be contacted by telephone to evaluate the status of their disease and to offer them, eventually, medical follow-up in our institution.

Ethics and Good Clinical Practices. The study protocol has been developed according to national standards for ethical, legal and juridical requirements, established in the Ministerial Resolution 1480/11 and international standards according to STROBE guidelines and according to ethical criteria of the Helsinki Declaration 2013, Nuremberg Code, Universal Declaration on Human Genome and Human Rights approved by the UNESCO General Conference 1997. As well as according to GCP standards (Good Clinical Practice). The confidentiality of all the data of each individual will be strictly maintained by means of the following strategies: the enrollment of the name, full ID and date of birth will be avoided, and will be replaced by coded data for the identification of the consequent methodologies according to this protocol.

Schedule of activities

* Medical records review phase: 6 months
* Phase of telephone calls: 3 months
* Results evaluation phase 3 months: end of the study and final variable measurements.

Expected results Describing, knowing, understanding the impact of the disease we expect to find a significant number of patients with chronic HCV who are lost to follow-up. Likewise, some of these patients will likely be in follow-up at other institutions.

ELIGIBILITY:
Inclusion Criteria:

* All of the following inclusion criteria must be met.
* Over 18 years old
* Diagnosis of chronic HCV

Exclusion Criteria:

* no

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCV viremic patients treatment naive or experienced
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
rate of relinked HCV patients | From Mayo 2024 to January 2025
  Strategy to re-engage HCV patients in a high complex hospital with a network of medium and low complexity hospitals.
proportion of relinked patients who received antiviral treatment | From Mayo 2024 to January 2025
  Strategy to re-engage HCV patients in a high complex hospital with a network of medium and low complexity hospitals.

SECONDARY OUTCOMES:
Evaluation and characteristics of the treatment established | From Mayo 2024 to January 2025
  * Describe the evolution of patients with HCV under follow-up.
  * describe the evolution and characteristics of HCV patients lost to follow-up.
  * Evaluate the number of patients relinked who effectively start treatment
  * Evaluate sustained virologic response rates and long-term clinical outcomes in patients who initiate treatment.
  * To evaluate SVR 4

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data underpinning the reported study results, including data used in analyses for text, tables, figures, and appendices, will be shared.
Supporting Information: Study Protocol
Time Frame: January 2025-January 2026
Access Criteria: Permission from the principal investigator is requested via email.
URL: https://www.hospitalelcruce.org/

REFERENCES:
- [Result] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. Lancet. 2007 Oct 20;370(9596):1453-7. doi: 10.1016/S0140-6736(07)61602-X. PMID 18064739
- [Result] Mendizabal M, Thompson M, Gonzalez-Ballerga E, Anders M, Castro-Narro GE, Pessoa MG, Cheinquer H, Mezzano G, Palazzo A, Ridruejo E, Descalzi V, Velarde-Ruiz Velasco JA, Marciano S, Munoz L, Schinoni MI, Poniachik J, Perazzo R, Cerda E, Fuster F, Varon A, Ruiz Garcia S, Soza A, Cabrera C, Gomez-Aldana AJ, Beltran FM, Gerona S, Cocozzella D, Bessone F, Hernandez N, Alonso C, Ferreiro M, Antinucci F, Torre A, Moutinho BD, Coelho Borges S, Gomez F, Murga MD, Pinero F, Sotera GF, Ocampo JA, Cortes Mollinedo VA, Simian D, Silva MO. Implementation of a re-linkage to care strategy in patients with chronic hepatitis C who were lost to follow-up in Latin America. J Viral Hepat. 2023 Jan;30(1):56-63. doi: 10.1111/jvh.13758. Epub 2022 Oct 17. PMID 36197907
- [Result] Wansom T, Falade-Nwulia O, Sutcliffe CG, Mehta SH, Moore RD, Thomas DL, Sulkowski MS. Barriers to Hepatitis C Virus (HCV) Treatment Initiation in Patients With Human Immunodeficiency Virus/HCV Coinfection: Lessons From the Interferon Era. Open Forum Infect Dis. 2017 Feb 11;4(1):ofx024. doi: 10.1093/ofid/ofx024. eCollection 2017 Winter. PMID 28480293
- [Result] Lazarus JV, Wiktor S, Colombo M, Thursz M; EASL International Liver Foundation. Micro-elimination - A path to global elimination of hepatitis C. J Hepatol. 2017 Oct;67(4):665-666. doi: 10.1016/j.jhep.2017.06.033. Epub 2017 Jul 29. No abstract available. PMID 28760329
- [Result] Mendizabal M, Alonso C, Silva MO. Overcoming barriers to hepatitis C elimination. Frontline Gastroenterol. 2019 Jul;10(3):207-209. doi: 10.1136/flgastro-2018-101114. Epub 2019 Feb 1. No abstract available. PMID 31288259
- [Result] Yehia BR, Schranz AJ, Umscheid CA, Lo Re V 3rd. The treatment cascade for chronic hepatitis C virus infection in the United States: a systematic review and meta-analysis. PLoS One. 2014 Jul 2;9(7):e101554. doi: 10.1371/journal.pone.0101554. eCollection 2014. PMID 24988388
- See also: Designing clinical reserch — https://edisciplinas.usp.br/pluginfile.php/5486505/mod_resource/content/1/Stephen%20B.%20Hulley%2C%20Steven%20R.%20Cummings%2C%20Warren%20S.%20Browner%2C%20Deborah%20G.%20Grady%2C%20Thomas%20B.%20Newm.pdf